CLINICAL TRIAL: NCT07291089
Title: Preoperative Pain-Risk Screening and Intervention for Intraoperative Pain in Second-Eye Cataract Surgery Based on Iris Vascular Area Density
Brief Title: Iris Vascular Area Density-Based Preoperative Pain-Risk Screening and Intervention in Second-Eye Cataract Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Huiyi Jin, Principal Investigator, Associate Chief Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCTR-2023C03-R
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Age Related Cataract; Pain Management During Cataract Surgery
Keywords: Cataract surgery; Pain; Second-eye cataract surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pranoprofen ophthalmic solution group (Experimental)
  Interventions: Drug: Pranoprofen eye drops
- Prednisolone acetate ophthalmic suspension group (Experimental)
  Interventions: Drug: Prednisolone acetate eye drops
- Sodium hyaluronate ophthalmic solution group (Placebo Comparator)
  Interventions: Drug: Sodium hyaluronate eye drops

INTERVENTIONS:
Drug: Pranoprofen eye drops — Participants receive one drop of pranoprofen instilled into the operative eye at 2 hours, 1.5 hours, 1 hour, and 30 minutes before cataract surgery.
  Arms: Pranoprofen ophthalmic solution group
Drug: Prednisolone acetate eye drops — Participants receive one drop of prednisolone acetate instilled into the operative eye at 2 hours, 1.5 hours, 1 hour, and 30 minutes before cataract surgery.
  Arms: Prednisolone acetate ophthalmic suspension group
Drug: Sodium hyaluronate eye drops — Participants receive one drop of sodium hyaluronate instilled into the operative eye at 2 hours, 1.5 hours, 1 hour, and 30 minutes before cataract surgery.
  Arms: Sodium hyaluronate ophthalmic solution group

SUMMARY:
This clinical trial aims to evaluate the effectiveness of pranoprofen or prednisolone acetate eye drops for pain management in patients undergoing second-eye surgery for age-related cataracts. Researchers will compare pranoprofen or prednisolone acetate eye drops with sodium hyaluronate eye drops to determine whether pranoprofen or prednisolone acetate eye drops can relieve intraoperative pain during second-eye cataract surgery.

Participants will:

1. Receive one drop in the operative eye at 2 hours, 1.5 hours, 1 hour, and 30 minutes before cataract surgery (pranoprofen, prednisolone acetate, or sodium hyaluronate)
2. Undergo cataract surgery and routine postoperative follow-up
3. Within 1 hour after surgery, provide a pain visual analog scale (VAS) score under the guidance of the investigator

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥50 years.
* Definite diagnosis of age-related cataract.
* The first-eye cataract surgery under local anesthesia has been completed at this hospital, and the second-eye cataract surgery under local anesthesia is planned with the same surgeon within 1 year of the first-eye surgery.
* Able to cooperate with preoperative iris optical coherence tomography angiography (OCTA) examination of the operative eye.
* On the day of the second-eye surgery, preoperative iris vascular area density (VAD) ≥ 0.2167 in the operative eye.

Exclusion Criteria:

* History of ocular trauma, ocular surgery (excluding the first-eye cataract surgery already performed), uveitis, chorioretinal disease, glaucoma;
* Presence of significant corneal disease, marked iris abnormalities, or any active ocular surface disease, including recent conjunctivitis, keratitis, or severe dry eye.
* Severe complications during or after the first-eye surgery (e.g., posterior capsule rupture, zonular dialysis, dislocation of the lens nucleus into the vitreous cavity, postoperative endophthalmitis, or glaucoma).
* History of chronic pain syndromes or neuropathic pain.
* Long-term use of opioids, other systemic analgesics, or sedative-hypnotic drugs.
* Known autoimmune disease or ongoing immunosuppressive therapy.
* Severe psychiatric disorders or cognitive impairment interfering with pain assessment.
* Use of topical corticosteroid eye drops in the second eye within 1 month prior to the planned surgery.
* Long-term use of α-adrenergic blockers or other medications associated with intraoperative floppy iris syndrome (IFIS).
* Participation in any other clinical trial involving ophthalmic or systemic drugs within the past 6 months.
* Known allergy or contraindication to topical nonsteroidal anti-inflammatory drugs (NSAIDs) (e.g., pranoprofen) or topical corticosteroids (e.g., prednisolone acetate) used in this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With Intraoperative Pain VAS ≥ 2 (Significant Pain) | Within 1 hour after surgery
  Intraoperative pain is assessed within 1 hour after surgery using a 0-10 visual analog scale (VAS; 0 = no pain, 10 = most severe pain). The investigator presents the unmarked side to the participant to mark perceived intraoperative pain; the investigator reads the corresponding value on the marked reverse side and records the score. The primary endpoint is the proportion of participants with VAS ≥ 2.

SECONDARY OUTCOMES:
Intraoperative Pain VAS Score | Within 1 hour after surgery
  VAS score on a 0-10 scale, obtained with the same standardized method as the primary outcome.
Patient-Reported Comparison of Second-Eye vs First-Eye Intraoperative Pain | Within 1 hour after surgery
  Within 1 hour after surgery, participants are asked to select one statement that best describes how pain during the second-eye surgery compares with their first-eye experience:
  1. "More painful than the first eye";
  2. "Less painful than the first eye";
  3. "About the same as the first eye";
  4. "I do not remember the pain during the first eye." The selected response is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu XJ, Wolff D, Zhang KK, He WW, Sun XH, Lu Y, Zhou P. Molecular Inflammation in the Contralateral Eye After Cataract Surgery in the First Eye. Invest Ophthalmol Vis Sci. 2015 Aug;56(9):5566-73. doi: 10.1167/iovs.15-16531. PMID 26305528
- [Background] Zhang Y, Du Y, Jiang Y, Zhu X, Lu Y. Effects of Pranoprofen on Aqueous Humor Monocyte Chemoattractant Protein-1 Level and Pain Relief During Second-Eye Cataract Surgery. Front Pharmacol. 2018 Jul 17;9:783. doi: 10.3389/fphar.2018.00783. eCollection 2018. PMID 30065652
- [Background] Cui L, Ma Y, Wang Y, Luo Q, Ding Q, Ge L, Lu S, Miao Y, Sun Q, Zou H, Jin H. Combination of iris vessel area density and surgery interval as the predictor of perceived pain during consecutive second-eye cataract surgery. J Cataract Refract Surg. 2023 Aug 1;49(8):858-863. doi: 10.1097/j.jcrs.0000000000001229. PMID 37350758